CLINICAL TRIAL: NCT05607433
Title: Air Q Intubating Laryngeal Airway (Air QILA) Versus the AmbuAura Gain as a Conduit for Endotracheal Intubation Assisted by Tube Exchanger, a Randomized Comparative Study.
Brief Title: Air Q Laryngeal Airway Versus the AmbuAura Gain as a Conduit for Endotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Zakaria Saleh Hassan Alrify, assistant lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: supraglottic devices
Record Dates: First submitted 2019-09-13; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Difficult Intubation
Keywords: assisted intubation

STUDY DESIGN:
Intervention Model Description: Randomized comparative study
Who Masked: Participant
Masking Description: only participants will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air Q ILA group (Experimental): Air Q supraglottic device will be placed in the participants in this group .
  Interventions: Device: cook ®Airway Exchanger Catheter
- Ambu AuraGain group (Experimental): Ambu AuraGain supraglottic device will be placed in the participants in this group .
  Interventions: Device: cook ®Airway Exchanger Catheter

INTERVENTIONS:
Device: cook ®Airway Exchanger Catheter — A tube exchanger is a small calibre , flexible tube used to guide endotracheal intubation through a supraglottic device.

SUMMARY:
The study aims to compare the efficacy of the Ambu AuraGain to that of the Air Q ILA as a conduit for endotracheal intubation assisted by tube exchanger. The comparison will be in terms of total intubation time, success rate of insertion of the tube exchanger as well as endotracheal intubation and complications.

DETAILED DESCRIPTION:
Very few studies discussed assisted endotrachealc intubation using certain tools as bougie through the Air Q ILA .

the hypothesis in this study is that the use of flexible, small calibre tube exchanger introduced through both supraglottic devices into the trachea as guidance for endotracheal intubation, will have shorter intubation time with the Ambu AuraGain than the Air Q ILA and less complications in both devices.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 60
* ASA physical status 1 and 2
* body weight less than 90 kilos
* Ganzouri airway score less than or equal to 3.

Exclusion Criteria:

* Active respiratory or cardiac disease
* Any expected airway difficulties
* Craniofacial abnormalities or fractures
* patients with abnormal coagulation profile

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Total endotracheal intubation time | time of tube exchanger insertion and endotracheal tube insertion
  tube exchanger intubation time plus endotracheal intubation time

SECONDARY OUTCOMES:
success rate of endotracheal intubation | 1 second after insertion tube exchanger until successful endotracheal intubation
  incidence of successful endotracheal intubation
Tube exchanger insertion time | from disconnection of the supraglottic device from ventilator to successful insertion of tube exchanger in trachea
  time from disconnection of the supraglottic device from ventilator to successful insertion of tube exchanger in trachea

OTHER OUTCOMES:
postoperative hoarseness of voice | 2 hours postoperative
  change of voice

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital, Cairo, Elmanial, Egypt

REFERENCES:
- [Background] Karim YM, Swanson DE. Comparison of blind tracheal intubation through the intubating laryngeal mask airway (LMA Fastrach) and the Air-Q. Anaesthesia. 2011 Mar;66(3):185-90. doi: 10.1111/j.1365-2044.2011.06625.x. PMID 21320087
- [Background] Bakker EJ, Valkenburg M, Galvin EM. Pilot study of the air-Q intubating laryngeal airway in clinical use. Anaesth Intensive Care. 2010 Mar;38(2):346-8. doi: 10.1177/0310057X1003800217. PMID 20369770